CLINICAL TRIAL: NCT06350292
Title: SLEEP-COPE: Sleep Enhancement and Effective Parenting for Children with Oppositional and Problematic Expressions
Brief Title: SLEEP-COPE: Sleep Intervention for Oppositional Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Melanie Stearns, Assistant Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0161464
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Insomnia Chronic; Oppositional Defiant Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Oppositional Defiant Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SLEEP: COPE (Experimental): Content includes both standard CBT-I techniques [sleep hygiene, stimulus control, sleep restriction, cognitive therapy] as well as those targeting children with ODD and their parents. Active child participation is a goal but may be limited due to age/abilities. Parents will work with children to implement behavioral strategies.
  Interventions: Behavioral: SLEEP: COPE

INTERVENTIONS:
Behavioral: SLEEP: COPE — Standard CBT-I techniques along with modules targeting noncompliance in children with ODD and their parents.

SUMMARY:
Children with Oppositional Defiant Disorder (ODD) are at risk for insomnia, arousal dysfunction, mood problems, and noncompliance. Cognitive behavioral treatment for insomnia (CBT-I) holds promise for improving insomnia and related concerns. Telehealth delivery will reduce the burden of in-person sessions, particularly in areas where there is low mental healthcare access. Telehealth CBT-I is efficacious in adults and children but has not been tested in children with ODD. The proposed trial is the next logical step - development and iterative testing of SLEEP-COPE, a brief dyadic telehealth CBT-I for children with ODD and their parents.

ELIGIBILITY:
Inclusion criteria:

1. Child ages 8-12 with ODD (prior diagnosis) and insomnia
2. Child and parent English proficiency.

Insomnia:

1. complaints of difficulties falling asleep, staying asleep, or early morning awakening by child report or parent observation for 3+ mos
2. daytime dysfunction (mood, cognitive, social, academic) due to insomnia
3. baseline diaries and actigraphy indicate >30 mins. of sleep onset latency, wake after sleep onset, or early morning awakening (time between last awakening and out of bed time) on 6+ nights

Exclusion criteria:

1. Parent unable to provide informed consent or child unable to provide assent
2. Family unwilling to accept random assignment
3. Child/parent participation in another randomized research project
4. Parent unable to complete forms or implement treatment procedures due to cognitive impairment
5. Child untreated medical comorbidity, including other sleep disorders (e.g., apnea, epilepsy, psychotic disorders, suicidal ideation/intent, [frequent] parasomnias)
6. Child psychotropic or other medications that alter sleep with the exceptions of stimulants, sleep medications, and/or melatonin
7. Child participation in non-pharmacological treatment (including CBT) for sleep outside current trial
8. Parent report of inability to undergo Holter Monitoring or actigraphy (e.g., extreme sensitivity, behavioral outbursts)
9. Other conditions adversely affecting trial participation

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Child Daily Sleep Diaries | Each morning for 14-days at 0 weeks, 6 weeks, and 10 weeks
  Daily diaries filled out by children with parent assistance that measure sleep efficiency, sleep onset latency, and total sleep time. Diaries also measure child behavior.
Parent Daily Sleep Diaries | Each morning for 14-days at 0 weeks, 6 weeks, and 10 weeks
  Daily diaries filled out by parents that measure sleep efficiency, sleep onset latency, and total sleep time. Diaries also measure parenting techniques.

SECONDARY OUTCOMES:
Child Actigraphy | 24/7 during the 2 week assessment at 0 weeks, 6 weeks, and 10 weeks
  Physiological measure of sleep efficiency, sleep onset latency, and total sleep time.
Parent Actigraphy | 24/7 during the 2 week assessment at 0 weeks, 6 weeks, and 10 weeks
  Physiological measure of sleep efficiency, sleep onset latency, and total sleep time.
Child Salivary Cortisol | before and after a cold-pressor task at 0 weeks, 6 weeks, 10 weeks
  Salivary cortisol collected in the morning before and after cold-pressor task and immediately frozen. Saliva samples (25 µL) assayed in duplicate. At rest children will undergo the following: 1) baseline saliva collection, 2) cold pressor stimulation to hand (place hand to bottom of 4° Celsius ice water) for 30 secs, 3) 3 min recovery, 4) cold pressor stimulation to other hand for 30secs, 5) post assessment saliva collection.
Child Hair Cortisol | 0 weeks, 6 weeks, 10 weeks
  Hair collected (15-50 mg) will be cut into 1 cm segments and ground into a fine powder before extracted with methanol for 16-18 hours while shaking. Cortisol then is quantified by liquid chromatography - tandem mass spectrometry (LC-MS/MS) (Salimetrics LLC, State College PA).
The Revised Childhood Anxiety and Depression Scale | 0 weeks, 6 weeks, 10 weeks
  Measures child anxiety and depression
PROMIS Child Sleep Disturbance | 0 weeks, 6 weeks, 10 weeks
  Measures child sleep
Alabama Parenting Questionnaire | 0 weeks, 6 weeks, 10 weeks
  Measures parenting behaviors
Perceived Stress Scale | 0 weeks, 6 weeks, 10 weeks
  Measures parent stress
Child Disruptive Behavior Disorders Checklist | 0 weeks, 6 weeks, 10 weeks
  Measures child disruptive behaviors
Beck Depression Inventory-II | 0 weeks, 6 weeks, 10 weeks
  Measures parent depression
State-Trait Anxiety Inventory | 0 weeks, 6 weeks, 10 weeks
  Measures parent anxiety
PROMIS Adult Sleep Disturbance | 0 weeks, 6 weeks, 10 weeks
  Measures parent sleep
Pediatric Sleep Questionnaire | 0 weeks, 6 weeks, 10 weeks
  Measures child sleep apnea risk
Epworth Sleepiness Scale | 0 weeks, 6 weeks, 10 weeks
  Measures parent sleep apnea risk

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No